CLINICAL TRIAL: NCT05607953
Title: A Phase 1/1b Pressure Enabled Regional Immuno-Oncology Study of Pancreatic Retrograde Venous Infusion of SD-101 Alone and With Checkpoint Blockade for Locally Advanced Pancreatic Ductal Adenocarcinoma
Brief Title: Pressure Enabled Intrapancreatic Delivery of SD-101 With Checkpoint Blockade for Locally Advanced Pancreatic Adenocarcinoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: TriSalus Life Sciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TS-PERIO-03
Record Dates: First submitted 2022-10-19; First posted 2022-11-07 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Locally Advanced Pancreatic Adenocarcinoma
MeSH Terms: interventions — spartalizumab

STUDY DESIGN:
Intervention Model Description: Phase 1: Two doses of SD-101 (given over two 52-day cycles) in dose-escalation fashion (0.5mg, 2mg, 4mg, 8mg-optional) via pancreatic retrograde infusion using pressure enabled drug delivery with the TriSalus Infusion System device.
  Phase 1b: Two doses of SD-101 (given over two 52-day cycles) at the maximum tolerated dose or optimal biologic dose defined in Phase 1b via pancreatic retrograde infusion using pressure enabled drug delivery with the TriSalus Infusion System device will be administered with systemic CPI.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- SD-101 (Experimental): Two doses of SD-101 given over two cycles via pancreatic retrograde venous infusion (PRVI) using the PEDD method of administration.
  Interventions: Drug: SD-101; Biological: anti-PD-1

INTERVENTIONS:
Drug: SD-101 — SD-101 doses are administered via PRVI using the PEDD method of administration
Biological: anti-PD-1 — In the Phase 1b, anti-PD-1 will be administered together with SD-101

SUMMARY:
This study is an open-label, phase 1/1b study of the pressure-enabled intrapancreatic infusion of SD-101, a TLR 9 agonist, alone or in combination with intravenous checkpoint blockade in adults with locally advanced pancreatic cancer.

DETAILED DESCRIPTION:
This study will be conducted in 2 phases.

In Phase 1, escalating doses of SD-101 will be administered alone via PRVI into the regional vessels of the pancreas containing the locally advanced tumor. The first three patients will part of a safety run-in. Following determination of the recommended MTD or optimal biologic dose (OBD) of SD-101 for PRVI, the study will progress to

Phase 1b to assess the safety of concomitant SD-101 and CPI usage, along with preliminary efficacy. Patients in Phase 1b will receive the SD-101 dose selected from Phase 1 together with systemic anti-PD-1, defined as any FDA approved anti-PD-1, checkpoint blockade. SD-101 will be administered over 2 cycles, with 1 dose per cycle and each cycle being about 6 weeks apart.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years of age with histologically or cytologically confirmed evaluable or measurable locally advanced unresectable PDAC, or previously confirmed disease in the absence of a documented complete pathologic response.
* Performance status score of 0 or 1 on the ECOG PS scale (scores range from 0 to 5, with higher numbers reflecting greater disability)
* Suitable venous anatomy on a standard portal venous phase imaging as defined by absence of portal, splenic, or superior mesenteric vein complete occlusion Note: As long as there is not complete occlusion and the Interventional Radiologist confirms that the target vein can be accessed, patients may be suitable for enrollment. All 3 veins do not have to be patent for eligibility.
* Having received standard of care chemoradiation therapy or a systemic chemotherapy regimen without a complete radiographic response. Standard of care chemotherapy includes gemcitabine + nab-paclitaxel, or FOLFIRINOX; for others discuss with medical monitor. Radiation with or without concurrent chemotherapy is also acceptable as a standard of care regimen
* Able to understand the study and provide written informed consent prior to any study procedures
* Has not received prior cytotoxic chemotherapy or targeted therapy within 14 days, or external radiation therapy within 4 weeks prior to screening
* Low-burden, asymptomatic metastatic disease permitted if:

  1. Metastatic disease poses no imminent threat to the patient
  2. Patient is otherwise asymptomatic with respect to metastases
  3. Metastases are limited to liver, lung, and/or bone
  4. No single lesion greater than 5 cm
  5. Less than 5 metastatic lesions total
  6. No brain or peritoneal metastases Pancreatic disease must be the dominant determinant of the patient's prognosis and clinical course
* Has no prior history of or other concurrent malignancy unless the malignancy is clinically insignificant, no ongoing treatment is required, and the patient is clinically stable
* Has a life expectancy of >3 months at screening as estimated by the Investigator
* Has a QTc interval ≤480 msec
* All associated clinically significant (in the judgment of the Investigator) drug-related toxicity from previous cancer therapy must be resolved (to Grade ≤1 or the patient's pretreatment level) prior to study treatment administration (Grade 2 alopecia, grade 2 peripheral neuropathy from prior chemotherapy, and endocrinopathies controlled on replacement therapy are allowed).
* Has adequate organ function at screening as evidence by:

  1. Platelet count >80,000/μL
  2. Hemoglobin ≥8.0 g/dL
  3. White blood cell (WBC) count >2,000/μL
  4. Serum creatinine ≤2.0 mg/dL unless the measured creatinine clearance is ≥30 mL/min calculated by Cockcroft-Gault formula.
  5. Total and direct bilirubin ≤2.0 × the upper limit of normal (ULN) and alkaline phosphatase ≤5 × ULN. For patients with documented Gilbert's disease, total bilirubin up to 3.0 mg/dL is allowed.
  6. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤5 × ULN
  7. Amylase and lipase ≤3 × ULN
  8. Prothrombin time/International Normalized Ratio (INR) or activated partial thromboplastin time (aPTT) test results at screening ≤1.5 × ULN (this applies only to patients who do not receive therapeutic anticoagulation; patients receiving therapeutic anticoagulation should be on a stable dose for at least 4 weeks prior to the first dose of study intervention) Note: Laboratory tests with exclusionary results judged by the Investigator as not compatible with the patient's clinical status may be repeated once for eligibility purposes.
* Females of childbearing potential must be nonpregnant and nonlactating, or post-menopausal, and have a negative serum human chorionic gonadotropin (hCG) pregnancy test result at screening and prior to the first dose of study intervention.

  1. Females of childbearing potential must agree to abstain from sexual activity with nonsterilized male partners, or if sexually active with a nonsterilized male partner must agree to use highly effective methods of contraception from screening, throughout the study and agree to continue using such precautions for 100 days after the final dose of study intervention.
  2. Nonsterilized males who are sexually active with a female of childbearing potential must agree to use effective methods of contraception and avoid sperm donation from Day 1 throughout the study and for 30 days after the final dose of study intervention.

Exclusion Criteria:

* Main portal, superior mesenteric vein, or splenic vein thrombosis with complete occlusion
* Severe portal hypertension, as evidenced by gastrointestinal (GI) bleeding, thrombocytopenia with splenomegaly
* Chronic pancreatitis
* Active autoimmune disease or history of IgG4 related pancreatitis
* Conversion to local resectability following prior treatment
* Has received chemotherapy or an investigational agent within 14 days (or 5 half-lives, whichever is shorter) before screening
* Has active, untreated brain metastasis
* Active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection
* Has main portal vein thrombosis, or severe portal hypertension as defined by a history of variceal hemorrhage or active ascites accumulation refractory to medical management
* Has Child-Pugh Class B or C cirrhosis.
* Has experienced a Grade 3 or higher immune-related AE from prior CPI therapy
* Is unable to be temporarily removed from chronic anticoagulation therapy
* Has a history of bleeding disorder
* Has active coronavirus disease 2019 (COVID-19), other severe infection, including a liver infection or acute pancreatitis, within 2 weeks before the first dose of study drug, or uncontrolled human immunodeficiency virus (HIV) infection at screening
* Has had bacterial pneumonia within 8 weeks of first dose of study drug
* Has active, known, or suspected autoimmune disease or immune-mediated disease. Type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis or alopecia) not requiring systemic treatment or conditions not expected to recur in the absences of an external trigger are not exclusionary
* Is receiving systemic steroid therapy >10 mg of prednisone daily or equivalent or any other immunosuppressive medication at any dose level. Local steroid therapies (e.g., otic, ophthalmic, intra-articular or inhaled medications) are acceptable
* Has significant concurrent or intercurrent illness, psychiatric disorder, or alcohol or chemical dependence that would, in the opinion of the Investigator and/or Medical Monitor, compromise their safety or compliance or interfere with interpretation of the study
* Lactating women are excluded from study participation
* Has previously received SD-101
* Medical history of significant hypersensitivity, severe and unresolved immune-mediated reactions, severe infusion-related reactions, or allergic reaction to TLR9 agonists or CPI agents in the judgment of the Investigator
* Patients who were enrolled in the Phase 1 portion of the study will not be eligible for enrollment in Phase 1b

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Phase 1 - To determine the maximum tolerated dose (MTD) or optimal biologic dose (OBD) of SD-101 administered alone via PRVI. | 12 months
  As a measure of safety, adverse events will be graded according to CTCAE v5.0
Phase 1b - To determine the safety of SD-101 administered via PRVI in combination with anti-PD-1 and to assess the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 disease control rate (DCR) | 12 months
  A standard 3+3 dose-escalation design will be employed to determine the MTD or optimal biologic dose.

SECONDARY OUTCOMES:
Phase 1 - To assess the RECIST v1.1 ORR | 12 months
  As a measure of activity, ORR will be assessed. ORR will be assessed using Response Evaluation Criteria in Solid Tumours (RECIST) v1.1.
Phase 1b - To assess the 12-month overall survival (OS) of PRVI of SD-101 in combination with intravenous (IV) immunological checkpoint blockade. | 12 months
  As a measure of activity, OS will be assessed. The events for the assessment of 12-month OS are death events.
Phase 1b - To assess preliminary efficacy in terms of RECIST for immune based therapeutics on ORR. | 12 months
  As a measure of activity, iRECIST will be utilized to determine overall response rate (ORR).
Phase 1b - To assess preliminary efficacy in terms of RECIST 1.1 pancreatic-specific response rate (PRR). | 12 months
  As a measure of activity, RECIST 1.1 will be utilized to determine pancreatic specific response rate.
Phase 1b - To assess preliminary efficacy in terms of RECIST 1.1 pancreatic-specific progression free survival (PPFS) | 12 months
  As a measure of activity, RECIST 1.1 will be utilized to determine pancreatic specific progression free survival
Phase 1b - To assess preliminary efficacy in terms of RECIST for immune based therapeutics on duration of response. | 12 months
  As a measure of activity, RECIST 1.1 will be utilized to determine duration of response (DOR)
Phase 1b - To assess preliminary efficacy in terms of RECIST for immune based therapeutics on clinical benefit ([CR] + [PR] + [SD]). | 12 months
  As a measure of activity, RECIST 1.1 will be utilized to determine clinical benefit (complete response [CR] + partial response [PR] + stable disease [SD]).
Phase 1b - To assess preliminary efficacy in terms of modified RECIST (mRECIST) for immune based therapeutics | 12 months
  As a measure of activity, mRECIST will be utilized to determine overall response rate (ORR).
Phase 1b - To assess preliminary efficacy in terms of RECIST 1.1 progression free survival (PFS) | 12 months
  As a measure of activity, RECIST 1.1 will be utilized to determine progression free survival (PFS)

CONTACTS AND LOCATIONS:
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States